CLINICAL TRIAL: NCT03670043
Title: Tolerance & Responsiveness Improvement for Metformin (TRIM): Open-label, Parallel-group Randomized Trial, Phase 4
Brief Title: Tolerance & Responsiveness Improvement for Metformin (TRIM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Side Institute for Science and Education (Other)
Responsible Party: Principal Investigator, Brian T. Layden, M.D., Ph.D., Chief, Section of Endocrinology, Jesse Brown VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1005965
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin ER (Active Comparator): The subjects developing GI-related symptoms with metformin will be randomized to Metformin Extended Release (ER)
  Interventions: Drug: Metformin Extended Release Oral Tablet
- Psyllium (Experimental): The subjects developing GI-related symptoms with metformin will be randomized to Psyllium
  Interventions: Drug: Psyllium powder

INTERVENTIONS:
Drug: Psyllium powder — To evaluate whether Psyllium will alleviate diarrhea
  Arms: Psyllium
Drug: Metformin Extended Release Oral Tablet — Metformin Extended Release Oral Tablet is standard of care for diarrhea in patients taking metformin
  Arms: Metformin ER

SUMMARY:
The overall goal is to explore the hypothesis that prebiotic fiber Psyllium will ameliorate diarrhea in African American men (AAM) with Type2 Diabetes Mellitus (T2D).

ELIGIBILITY:
Inclusion criteria

1. Male (M)
2. African American (AA) race
3. Age 20-70 years
4. BMI 28-59 kg/m2
5. T2D
6. A1c 6.5 - 8.9%
7. eGFR =/> 30
8. Drug-naïve or use Glipizide or newly started on Metformin (within 2 weeks).

Exclusion criteria

1. Chronic kidney disease stage 3b, 4 and 5 (eGFR < 30)
2. Insulin use
3. Oral steroids use (inhalers and creams are allowed)
4. Antibiotic use within the last month
5. Artificial heart valves
6. Hospitalization for chronic condition within 6 months prior to the study
7. History, manifestations or medications of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, psychiatric/ psychological disorders, or social circumstances which in the opinion of the investigator would be expected to interfere with the study or increase risk to the subject.
8. Use of other antidiabetic drugs (except glipizide and metformin).
9. Acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma.

Additional Exclusion criteria for subjects who previously used Metformin:

1. Previous severe allergic reaction to metformin hydrochloride, such as angioedema.
2. Previous Metformin intolerance causing significant diarrhea or GI-upset. Would not exclude participants who had history of mild diarrhea with metformin use.
3. Previous side effects that the subject feels were related to Metformin and the subject is not interested to re-try metformin.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Birmingham Irritable Bowel Syndrome (IBS) Symptom Questionnaire | 3 months
  This scale is based on symptoms that frequently occur in IBS cases, examines abdominal discomfort status, stool properties, and defecation feelings. The scale includes a total of 11 items, with 6 possible grades for each item that range from 0 points (never having this symptom) to 5 points (the symptom is always present). The total score is the sum of the scores for each item. The Total score is used. No "subscale" is used. Total range is minimum=0, maximum=55. The higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Barengolts, Principal Investigator — Jesse Brown VA Medical Center
Locations (1):
- Jesse Brown VA Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT03670043/ICF_000.pdf